CLINICAL TRIAL: NCT02609594
Title: A Multi-center Randomized Controlled Clinical Trial Evaluating Two Application Regimens of Amnioband Dehydrated Human Amniotic Membrane and Standard of Care vs. Standard of Care Alone in the Treatment of Venous Leg Ulcers
Brief Title: Amnioband and Standard of Care vs. Standard of Care Alone in the Treatment of Venous Leg Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SerenaGroup, Inc. (Network)
Collaborators: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Principal Investigator, Thomas Serena, Principal Investigator, SerenaGroup, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMNIOVLU01
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Venous Leg Ulcers
Keywords: human amniotic membrane; compression therapy; venous leg ulcer
MeSH Terms: conditions — Varicose Ulcer | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard of Care (Active Comparator): Subjects randomized to this group will receive standard of care (multi-layer compression therapy).
  Interventions: Other: Standard of Care
- Weekly application of Amnioband (Experimental): Weekly application of Amnioband plus standard of care.
  Interventions: Other: Weekly application of Amnioband; Other: Standard of Care
- Biweekly application of Amnioband (Experimental): Biweekly application of Amnioband plus standard of care.
  Interventions: Other: Biweekly application of Amnioband; Other: Standard of Care

INTERVENTIONS:
Other: Weekly application of Amnioband — Weekly application of Amnioband.
  Arms: Weekly application of Amnioband
Other: Biweekly application of Amnioband — Biweekly application (every two weeks) of Amnioband.
  Arms: Biweekly application of Amnioband
Other: Standard of Care — Standard of care for this study is weekly multi-layer compression bandaging.

SUMMARY:
Lower extremity ulcers pose significant clinical, humanistic and economic burdens on society. Millions of Americans are afflicted with painful, open, draining sores on their lower extremities. These sores are referred to as venous leg ulcerations (VLUs).1-5 Under the best of circumstances these ulcers require weeks or months to heal. Not uncommonly wound care specialists see patients who have suffered for years or faced amputation of the limb as their only option to alleviate the pain.

Standard of care will result in healing in 50% of venous leg ulcers in 12 weeks. However, roughly half of patients suffering from venous ulcers will require advanced therapy. Human amniotic membrane replaces the damaged extracellular matrix characteristic of chronic ulcers. In addition, it contains cytokines that may accelerate healing. In clinical practice and recent studies, Dehydrated Human Amniotic Membrane has appeared to be as effective as bioengineered skin products. This RCT is designed to evaluate Amnioband Dehydrated Human Amniotic Membrane in venous leg ulcers.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, trial designed to evaluate the safety and effectiveness of Amnioband Dehydrated Human Amniotic Membrane plus multi-layer compression therapy versus multi-layer compression alone in the healing of venous leg ulcers.

The Standard of Care therapy in this study is multi-layer compression therapy. A number of compression bandaging systems are commercially available. The choice of compression will be at the discretion of the principle investigator.

The Screening Phase (1-14 days) consists of a series of screening assessments designed to determine eligibility followed by, for those who meet the eligibility criteria (described in more detail below), At or up to 14 days before the first Screening Period Visit (S1), written informed consent from the subject will be obtained by the Investigator or suitably qualified designee before the performance of any other protocol-specific procedure.

Subjects who have not been treated with compression therapy for the target ulcer must receive a minimum of 14 days of compression prior to enrollment.

At the first Screening Period Visit (S1), the Investigator will select the study (target) ulcer. Each subject will have only one VLU selected as the study (target) ulcer. In the situation where a subject has more than one VLU at the S1 visit, the Investigator will select the largest VLU that meets the eligibility criteria of the protocol as the study (target) ulcer.

The Screening Period is designed to determine whether subjects are eligible to proceed to the Treatment Period of the study.

The Treatment Phase (12 Weeks) begins with a series of assessments designed to confirm the subjects' continued eligibility. Subjects who continue to meet eligibility criteria will be randomized to one of three groups: (1) standard of care: multi-layer compression (2) weekly application of Amnioband Dehydrated Human Amniotic Membrane (3) biweekly applications of Amnioband Dehydrated Human Amniotic Membrane.

During the Treatment Phase, subjects will be evaluated on a weekly basis. Efficacy evaluations each week will include Investigator assessment of ulcer healing and measurements of ulcer size using a digital camera device. Safety evaluations during the Treatment Phase will consist of adverse event assessments at each visit.

Subjects in any of the three groups whose ulcers do not achieve closure at 12 weeks will be deemed treatment failures. Subjects in the control arm may cross over to the Amnioband arm if they fail to achieve closure although these subjects will not be included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Ankle Brachial Pressure Index (ABI) > 0.75 OR SPP > 30 mmHg OR TCOM > 30 mmHg.*
3. Presence of a venous leg ulcer extending through the full thickness of the skin but not down to muscle, tendon or bone.
4. The largest ulcer will be designated the index ulcer and the only one included in the study. If other ulcerations are present on the same leg they have to be more than 2 cm apart from the index ulcer.
5. Study ulcer (i.e. current episode of ulceration) has been present for greater than one month prior to the initial screening visit, and has failed to respond to documented conservative measures for greater than (1) one month duration and is excluded if it has undergone 12 months of continuous high strength compression therapy over its duration.
6. Study ulcer is a minimum of 2 cm2 and a maximum of 20 cm2 at the randomization visit.
7. The target ulcer has been treated with compression therapy for at least 14 days prior to randomization.
8. Ulcer has a clean, granulating base with minimal adherent slough at the randomization visit.
9. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence).
10. Subject understands and is willing to participate in the clinical study and can comply with weekly visits and the follow-up regimen.
11. Subject has read and signed the IRB/IEC approved Informed Consent Form before screening procedures are undertaken.

Exclusion Criteria:

1. Study ulcer(s) deemed by the investigator to be caused by a medical condition other than venous insufficiency.
2. Study ulcer exhibits clinical signs and symptoms of infection.
3. Known allergy to the components of the multi-layer compression bandaging, or who cannot tolerate multi-layer compression therapy.
4. Study ulcer, in the opinion of the investigator, is suspicious for cancer should undergo an ulcer biopsy to rule out a carcinoma of the ulcer.
5. Subjects with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within one month prior to initial screening, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
6. Subjects on any investigational drug(s) or therapeutic device(s) within 30 days preceding Screening.
7. Study ulcer improving greater than 30% during the screening phase if the subject was not in adequate compression 14 days prior to screening.
8. History of drug or alcohol abuse.
9. History of radiation at the ulcer site.
10. Presence of one or more medical conditions, as determined by medical history, hematologic, active auto-immune or immune diseases that, in the opinion of the Investigator, would make the subject an inappropriate candidate for this ulcer healing study.
11. History of having Acquired Immunodeficiency Syndrome (AIDS) or HIV.
12. Study ulcer has been previously treated with tissue engineered materials (e.g. Apligraf® or Dermagraft®) or other scaffold materials (e.g. Oasis, Matristem) within the last 30 days
13. Study ulcer requiring negative pressure wound therapy or hyperbaric oxygen during the course of the trial.
14. Presence of any condition(s) which seriously compromises the subject's ability to complete this study, or has a known history of poor adherence with medical treatment.
15. Ulcers on the dorsum of the foot or with more than 50% of the ulcer below the malleolus are excluded.
16. Pregnant or breast feeding.
17. Presence of diabetes with poor metabolic control as documented with a HgA1c > 12.0 within last 90 days
18. Patients with renal dysfunction whose serum creatinine levels are 3.0mg/dl or greater within the last 90 days
19. History of usage of tobacco products within the last 30 days
20. History of Liver disease with active Cirrhosis of the liver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Time to complete ulcer closure | 12 weeks
  Ulcer closure is based on wound area measurement and absence of wound exudate.

SECONDARY OUTCOMES:
Proportion of ulcers achieving 40% ulcer closure | 4 weeks
  This is measured by wound area.
Percentage of ulcers achieving complete closure | 12 weeks
  This is measured by wound area and absence of wound exudate.
Incidence of adverse events | 12 weeks
Cost effectiveness | 12 weeks
  The per unit cost of providing wound care is known. The use of amniotic membrane to standard of care will be compared in terms of the cost of achieving healing.
Reduction in pain between treatment groups | 12 weeks
  Pain is measured by subject report on a scale of 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Squillante, Study Director — Musculoskeletal Transplant Foundation
Locations (8):
- United States (8):
  - Brigham and Women's Hospital Wound Care Center, Boston, Massachusetts
  - Premier Surgical, Brick, New Jersey
  - Inspira Medical Center - Elmer Wound Care Center, Elmer, New Jersey
  - St John Medical Center, Tulsa, Oklahoma
  - The Foot and Ankle Wellness Center, Ford City, Pennsylvania
  - Armstrong County Memorial Hospital, Kittanning, Pennsylvania
  - SerenaGroup Research Institute, Pittsburgh, Pennsylvania
  - Martinsville Research Institute, Martinsville, Virginia